CLINICAL TRIAL: NCT03471494
Title: GlobalSurg 3: Quality and Outcomes in Global Cancer Surgery
Acronym: GS3
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: GS3
Record Dates: First submitted 2018-03-09; First posted 2018-03-20 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms; Gastric Cancer; Colon Cancer
Keywords: Surgery; Quality; Outcomes
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer
  Interventions: Other: Exposure: human development index of country
- Gastric cancer
  Interventions: Other: Exposure: human development index of country
- Colon cancer
  Interventions: Other: Exposure: human development index of country

INTERVENTIONS:
Other: Exposure: human development index of country — Primary comparison: Between country groups defined by human development index.

SUMMARY:
Aim The aim is to determine the variation in quality of cancer surgery worldwide. Quality will be determined using measures covering infrastructure, care processes, and outcomes. The study will concentrate on the most common surgically treated cancers worldwide: breast, gastric and colorectal cancer. The primary aim focusses on 30-day mortality and complication rates after cancer surgery. The secondary aim is to characterise infrastructure and care processes in the treatment of these cancers worldwide.

Primary outcome measure 30-day mortality and complication rates after cancer surgery.

Primary comparison Between country groups defined by human development index.

Hospital eligibility Any hospital in the world performing surgery for breast, gastric or colorectal cancer.

Patient eligibility Consecutive patients undergoing surgery for breast, gastric, or colorectal cancer. Surgery can be with palliative or curative intent.

Team Individual hospital teams with up to three people, collecting data for four weeks. Several teams collecting data over multiple four-week periods is encouraged.

Time period Patients will be identified, and data collected on all patients during the time-period with follow-up to 30-days. The study will run from 1st April 2018 to 31st October 2018 (with follow-up of the last period to 30th November 2018).

Validation Data validation will be in two parts. First, centres will self-report the key processes used to identify and follow-up patients. Second, independent validators will quantitatively report case ascertainment and sampled data accuracy.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing therapeutic surgery (curative or palliative) for breast, gastric, and colorectal cancer should be included.
* Surgery is defined as a procedure requiring a skin incision performed under general or neuraxial (e.g. regional, epidural or spinal) anaesthesia.
* Both elective and emergency procedures should be included. Include patients in whom the pre-operative diagnosis was thought to be benign, but was subsequently found to be cancer, e.g. bowel obstruction found to be due to cancer during surgery.
* Include patients in whom the pre-operative diagnosis was thought to be cancer, but was subsequently found to be benign disease (ensure the "pathology" variable indicates not cancer; will not be included in primary analysis).
* Laparoscopic, laparoscopic-converted, robotic, and open cases should be included.
* Patients aged 18 years and over should be included .
* Surgery may be with curative or palliative intent. Include patients in whom curative surgery was attempted but abandoned, e.g. open/close laparotomy.

Exclusion Criteria:

* Operations where breast, gastric, or colorectal cancer is not suspected to be the primary pathology should be excluded.
* Patients undergoing a procedure purely for diagnosis or staging should be excluded, e.g. open breast biopsy, staging laparoscopy.
* Patients undergoing a procedure which does not require a skin incision should be excluded, e.g. colonoscopy/endoscopy alone, chemo/radiotherapy alone.
* Patients presenting with recurrence of breast, colorectal or gastric cancer should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective or emergency surgery for breast, gastric, or colorectal cancer anywhere in the world are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 15958 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate | 30 days from surgery
  Death within 30 days of surgical procedure
30-day complication rate | 30 days from surgery
  Defined with by Clavien-Dindo grade III or IV

SECONDARY OUTCOMES:
Availability/performance of pre-operative fine needle aspiration/core biopsy to diagnose breast cancer. | Prior to surgery.
  For breast cancer.
Availability/performance of breast/axillary MRI for staging. | Prior to surgery.
  For breast cancer.
Availability/performance of breast conservation surgery for AJCC stage 0/I/II breast cancer. | Prior to surgery.
  For breast cancer.
Availability/ performance of axillary/breast radiotherapy and axillary lymph node clearance. | Collection of variable within 30 days of surgery.
  For breast cancer.
Availability/performance of sentinel lymph-node biopsy for early invasive breast cancer. | During surgery.
  For breast cancer.
Availability/performance of progesterone receptor (PR), oestrogen receptor (ER), human epidermal growth factor receptor 2 (HER2) receptor and Ki67 status for invasive cancers. | Prior to surgery.
  For breast cancer.
Availability/treatment with adjuvant treatment where appropriate within 31 days of completion of surgery. | Within 31 days of completion of surgery.
  For breast cancer.
Availability/plan for radiotherapy for all with breast conserving surgery with clear margins (including DCIS). | Collection of variable within 30 days of surgery.
  For breast cancer.
Margin involvement. "Tumour on inked margin" is considered positive (SSO/ASTRO consensus guidelines) in surgery for early stage breast cancer or a margin <2 mm in DCIS [or ability to measure this locally]. | Collection of variable within 30 days of surgery.
  For breast cancer.
Availability/performance of CT chest, abdomen and pelvis scan performed for pre-operative staging. | Prior to surgery.
  For gastric cancer.
Availability/treatment with pre- or post-operative chemotherapy for gastric cancer. | Prior to surgery.
  For gastric cancer.
Treatment decisions made within multidisciplinary team meeting / tumour board. | Prior to surgery.
  For gastric cancer.
At least 15 regional lymph nodes removed and pathologically examined for resected gastric cancer [or ability to measure this locally]. | Collection of variable within 30 days of surgery.
  For gastric cancer.
Availability/performance of CT chest, abdomen and pelvis scan performed for pre-operative staging. | Prior to surgery.
  For colon cancer.
Availability/performance of pre-operative MRI for rectal cancer. | Prior to surgery.
  For colon cancer.
Availability/planning/treatment with post-operative chemotherapy following resection for lymph node positive colon cancer. | Collection of variable within 30 days of surgery.
  For colon cancer.
Availability/treatment with pre-operative chemotherapy/radiotherapy. | Prior to surgery.
  For colon cancer.
Treatment decisions made within multidisciplinary team meeting / tumour board. | Prior to surgery.
  For colon cancer.
Stoma formation rate. | During surgery.
  For colon cancer.
Circumferential resection margin (CRM) >1mm [or ability to measure this locally]. | Collection of variable within 30 days of surgery.
  For colon cancer.
At least 12 regional lymph nodes removed and pathologically examined for resected colon cancer [or ability to measure this locally]. | Collection of variable within 30 days of surgery.
  For colon cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Derived anonymised data at the patient-level may be able to be made available for sharing.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] GlobalSurg Collaborative and National Institute for Health Research Global Health Research Unit on Global Surgery. Global variation in postoperative mortality and complications after cancer surgery: a multicentre, prospective cohort study in 82 countries. Lancet. 2021 Jan 30;397(10272):387-397. doi: 10.1016/S0140-6736(21)00001-5. Epub 2021 Jan 21. PMID 33485461
- [Derived] NIHR Global Health Research Uniton Global Surgery. Quality and outcomes in global cancer surgery: protocol for a multicentre, international, prospective cohort study (GlobalSurg 3). BMJ Open. 2019 May 24;9(5):e026646. doi: 10.1136/bmjopen-2018-026646. PMID 31129582
- See also: Related Info — http://globalsurg.org/gs3